CLINICAL TRIAL: NCT04860960
Title: Phase 3, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of 2000mg/kg of Trappsol®Cyclo™ (Hydroxypropyl-B-cyclodextrin) and Standard of Care Compared to Placebo and Standard of Care in Patients With Niemann-Pick Disease Type C1 (TransportNPC)
Brief Title: Phase 3 Study to Evaluate Intravenous Trappsol(R) Cyclo(TM) in Pediatric and Adult Patients With Niemann-Pick Disease Type C1
Acronym: TransportNPC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cyclo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTD-TCNPC-301
Record Dates: First submitted 2021-04-15; First posted 2021-04-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-09

CONDITIONS: Niemann-Pick Disease, Type C1
Keywords: NPC1; cyclodextrin; Niemann-Pick; Niemann-Pick Type C; NPC; Niemann Pick C; Niemann Pick Type C; Niemann Pick
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, multi-center, double-blind and parallel group study with 2:1 randomization of Trappsol Cyclo plus SOC versus placebo plus SOC over 96 weeks, followed by open-label extension study of 96 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Intravenous administration of 2000 mg/kg hydroxypropyl betacyclodextrin (Trappsol Cyclo) (based on body weight) diluted with 0.5N saline over at least 6.5 hours every 2 weeks
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin
- Placebo comparator (Placebo Comparator): Intravenous administration of 0.5N saline over at least 6.5 hours every 2 weeks
  Interventions: Drug: Placebo
- Open Label sub-study for Infants up to age 3 (Experimental): Up to 12 patients age 0 - 3 yrs in countries following EMA guidance may be enrolled in this open label sub-study. All patients will receive 2000 mg/kg hydroxypropyl betacyclodextrin (Trappsol Cyclo) diluted with 0.5N saline at the clinician's discretion over 6.5 hours every 2 weeks. Outcome measures are safety, clinician and caregiver impressions.
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin

INTERVENTIONS:
Drug: Hydroxypropyl-beta-cyclodextrin — Dose is 2000 mg/kg body weight provided every 2 weeks intravenously
  Other Names: Trappsol Cyclo
  Arms: Experimental; Open Label sub-study for Infants up to age 3
Drug: Placebo — 0.5N saline provided every 2 weeks intravenously
  Other Names: 0.5N saline
  Arms: Placebo comparator

SUMMARY:
A prospective, randomized, double-blind, placebo controlled, multi-center therapeutic study for patients age 3 and older with confirmed diagnosis of Niemann Pick disease type C1 (NPC1). The objective of this study is to evaluate the safety, tolerability and efficacy of 2000 mg/kg dose of Trappsol Cyclo (hydroxypropyl betacyclodextrin) administered intravenously compared to standard of care. An open-label sub-study in countries following European Medicines Agency (EMA) guidance will enroll asymptomatic or symptomatic patients from infancy up to age 3 to evaluate safety in that population.

DETAILED DESCRIPTION:
The TransportNPC study is a prospective, randomized, double-blind, placebo controlled therapeutic study for 93 patients age 3 and older with confirmed diagnosis of NPC1. The objective of this study is to evaluate the safety, tolerability and efficacy of 2000 mg/kg dose of Trappsol Cyclo (hydroxypropyl betacyclodextrin) administered intravenously by slow infusion every two weeks in addition to standard of care as compared to placebo and standard of care. Standard of care may include Miglustat or leucine products that are not currently under investigation as a therapeutic. Patients will be randomized to receive Trappsol Cyclo or placebo at a 2:1 ratio. The study duration is 96 weeks, with an unblinded interim analysis at 48 weeks. An open-label extension of up to 96 weeks follows the interventional study. Patients whose disease progression worsens by two levels in the Clinical Global Impression of Severity scale over 12 weeks, starting at week 36, may be moved to open label treatment. Efficacy will be measured at week 48 and week 96 by a composite score of major disease features. A sub-study will be conducted in countries following EMA guidance for up to 12 patients age 0 - 3 years who may be asymptomatic. Outcomes for the sub-study are safety, clinical and caregiver impression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of NPC1
2. Annual Severity Increment Score between 0.5 and 2.0 using the 17-domain NPC Severity Scale
3. Treated or Not Treated with Miglustat (patients must be on a stable dose for at least 3 months prior to the Screening Visit, or have discontinued Miglustat for at least 3 months prior to Screening Visit).
4. Body weight greater than 4.5 kg and less than or equal to 125 kg
5. Presenting at least 1 neurological symptom of the disease
6. Written informed consent
7. Willing and capable to participate in all aspects of trial design
8. Ability to travel to the trial site at scheduled times
9. Contraception requirements per protocol
10. Caregiver consent as appropriate to participate in all protocol-specified assessments for duration of trial
11. Inclusion criteria for Open Label Extension are 1) Received double-blind treatment for at least 48 weeks with CGI-S deterioration by at least 2 levels for 2 consecutive assessment visits 12 weeks apart, or 2) completion of double-blind treatment and completed all assessments through week 96, or 3) Discontinued early from double-blind treatment but completed all assessments through week 96
12. Inclusion criteria for patients age 0 to 3 years in open-label sub-study in countries following EMA guidance only: Confirmed diagnosis of NPC1; treated or not with Miglustat per main study; body weight greater than 4.5kg; patient may be asymptomatic; written assent for child to participate in safety assessments; caregiver consent to participate in caregiver assessments; ability to travel to the trial site for all scheduled visits.

Exclusion Criteria:

1. Recipient of a liver transplant within <12 months or planned liver transplantation
2. Patients with active liver disease from any cause other than NPC1
3. Clinical evidence of acute liver disease including symptoms of jaundice or right upper quadrant pain or international normalized ratio > 1.8
4. Stage 3 chronic kidney disease or worse as indicated by an estimated glomerular filtration rate <60ml/min/1.73m2.
5. Use of curcumin or fish oil within 12 weeks prior to enrollment
6. Known or suspected allergy or intolerance to the study treatment
7. In the opinion of the Investigator, the patient's clinical condition does not allow for the blood collection required as per protocol specific procedures.
8. Treatment with any investigational drug during the 3 months prior to entering the study. If the investigational drug has a short half-life (<8 hours) and would be expected to be cleared from the body within 1 month, then the wash-out period is 1 month. Treatment with any form of leucine, whether as an investigational drug or other formulation is not allowed
9. Treatment with any other investigational drug during the study
10. Pregnancy or breastfeeding
11. Current participation in another trial is not permitted unless it is a noninterventional study and the sole purpose of the trial is for long-term follow up describing clinical features or survival data (registry)
12. Patients with uncontrolled, severe epileptic seizure periods (at least 3 consecutive severe epileptic seizures that required medication) within 2 months prior to completion of informed consent or assent, as applicable.
13. Neurologically asymptomatic patients
14. Inability to participate in the primary study assessment (4D-NPC-SS or 5D-NPC-SS) as determined by the Investigator
15. Exclusion criteria for patients age 0 to 3 years in open-label sub-study in countries following EMA guidance only are similar to the main study with the addition of exclusion criterion of history of fetal hydrops or fetal ascites

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 4-Domain NPC Severity Score (US only) | Interim Analysis at Week 48
  Ambulation, Fine Motor, Speech, Swallow
Change from Baseline in 4-Domain NPC Severity Score (US only) | End of Study at Week 96
  Ambulation, Fine Motor, Speech, Swallow
Change from Baseline in 5-Domain NPC Severity Score (ex-US) | Interim Analysis at Week 48
  Ambulation, Fine Motor, Speech, Swallow, Cognition
Change from Baseline in 5-Domain NPC Severity Score (ex-US) | End of Study at Week 96
  Ambulation, Fine Motor, Speech, Swallow, Cognition

SECONDARY OUTCOMES:
Change in ataxia as measured by Spinocerebellar ataxia functional index | Change from Baseline as measured every 12 weeks through week 96 and end of OLE week 192
  SCAFI
Change in adaptive behavior as measured by Vineland Adaptive Behavior Scale II | Change from Baseline as measured every 12 weeks through week 96 and end of OLE week 192
  Vineland Adaptive Behavior Scale II
Change in Swallow function evaluated by videofluoroscopy or fiberoptic endoscopy and measured by Penetration Aspiration Scale | Change from Baseline measured at Interim Analysis Week 48
  PAS
Change in Swallow function evaluated by videofluoroscopy or fiberoptic endoscopy and measured by Penetration Aspiration Scale | Change from Baseline measured at End of Study Week 96
  PAS

OTHER OUTCOMES:
Change in speaking ability compared to Baseline as measured by voice recordings collected in SpeechVitals mobile device application | Baseline and every two weeks through week 192
  Measurement of speech features including articulatory precision, speaking and pause rates
Change in speaking ability compared to Pre-Infusion as measured by voice recordings collected in SpeechVitals mobile device application | Every two weeks through week 192
  Measurement of speech features including articulatory precision, speaking and pause rates within 24 hours post-infusion
Change in Scores of Clinical Global Impression of Severity and of Change compared to Baseline | Baseline, weeks 2, 4, 12, 24, 36, 48, 60, 72, 84, 96, 100, 120, 144, 168, 192
  Clinical Global Impression of Severity and of Change
Change in Scores of Caregiver Global Impression of Severity and of Change scales | Baseline, weeks 2, 4, 12, 24, 36, 48, 60, 72, 84, 96, 100, 120, 144, 168, 192
  Caregiver Global Impression of Severity and of Change
Caregiver Global Impression of Change at 24 hours post infusion | Baseline and every 2 weeks through week 192
  Caregiver Global Impression of Change at 24 hours post infusion
Change from Baseline in Respiratory function measured by Forced Expiratory Volume in 1 second | Baseline, weeks 2, 4, 12, 24, 36, 48, 60, 72, 84, 96, 100, 192
  FEV1
Change from Baseline in Liver function as measured by liver enzyme assessments | Baseline, weeks 2, 4, 12, 24, 36, 48, 60, 72, 84, 96, 100, 120, 144, 168, 192
  Liver function measured by liver enzyme assessments including alanine and aspartate aminotransferases
Safety assessments to include incidence of Adverse Events and Serious Adverse Events | Regular assessments per protocol through week 192
  Incidence of AEs, SAEs, incidence of abnormal laboratory test results, abnormal ECGs, abnormal physical exams, abnormal vital signs and abnormal hearing assessments assessments

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mullen, MD, Study Director — Cyclo Therapeutics, Inc.
Locations (35):
- United States (7):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Florida, Jacksonville, Florida
  - Emory, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Children's Hospital, Pittsburgh, Pennsylvania
  - University Utah, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research & Treatment Center, Inc., Fairfax, Virginia
- Argentina (2):
  - Hospital de Alta Complejidad en Red "El Cruce", Buenos Aires
  - Hospital de Niños de la Santísima Trinidad, Córdoba
- Australia (3):
  - Melbourne Children's Trials Centre Murdoch Children's Research Institute, Parkville, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Metabolic Clinical Trials Unit, Adelaide
- Brazil (3):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Universidade de São Paulo, São Paulo
  - University of Campinas, São Paulo
- Germany (2):
  - SphinCS GmbH, Höchheim
  - University Munster, Münster
- Israel (2):
  - Emek Medical Center-Department of Pediatrics, Afula
  - Soroka Medical Center, Beersheba
- Italy (4):
  - University of Catania, Catania
  - Istituto Neurologico Carlo Besta, Milan
  - University Hospital of Padova, Padua
  - Centro di Coordinamento Regionale Malattie Rare, Udine
- Poland (2):
  - Szpital Uniwersytecki w Krakowie, Krakow
  - MediPark, Warsaw
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- Spain (3):
  - Hospital Sant Joan de Déu - Neurology Department, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- National Taiwan University Hospital, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Gazi University Faculty of Medicine, Ankara
  - Ege University Medical School, Department of Inborn Errors of Metabolism, Izmir
- United Kingdom (3):
  - Birmingham Children's Hospital NHS Foundation Trust · Department of Inherited Metabolic Disorders Service, Birmingham
  - University College London, London
  - Salford Royal Foundation NHS Trust, Salford

REFERENCES:
- [Derived] Hastings C, Liu B, Hurst B, Cox GF, Hrynkow S. Intravenous 2-hydroxypropyl-beta-cyclodextrin (Trappsol(R) Cyclo) demonstrates biological activity and impacts cholesterol metabolism in the central nervous system and peripheral tissues in adult subjects with Niemann-Pick Disease Type C1: Results of a phase 1 trial. Mol Genet Metab. 2022 Dec;137(4):309-319. doi: 10.1016/j.ymgme.2022.10.004. Epub 2022 Oct 17. PMID 36279795